CLINICAL TRIAL: NCT00164073
Title: Pharmacogenomics of Interferon and Ribavirin Treatment in Patients With Chronic Hepatitis C Virus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: University of Adelaide (Other)
Other Study IDs: 122/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis C
Keywords: HCV and microarray; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Liver biopsy

SUMMARY:
The purpose of this study is to examine gene expression profiles by DNA microarray in patients who are responders and non-responders to interferon and ribavirin treatment for hepatitis C virus (HCV). Genes involved in inflammation and fibrosis and mediators of the Th-1 lymphocyte response will be looked for. It is hoped that genetic targets for future more effective and less toxic treatments will be identified.

DETAILED DESCRIPTION:
Background and Research Plan:

Chronic HCV infection often follows a progressive course over many years, and can ultimately result in cirrhosis and the need for liver transplantation or hepatocellular carcinoma. The decision to treat patients with chronic hepatitis C infection is based upon several factors including the natural history and stage of the disease and the efficacy and adverse effects related to therapy. As a general rule patients who are considered for treatment should have histologic and virologic evidence of chronic infection (i.e., HCV RNA detectable in serum) and an elevated serum ALT (1). Combination treatment with Interferon and Ribavirin is currently the best available treatment for chronic HCV infection. However, response to therapy is suboptimal and there are several side effects.

Side effects seen during therapy of patients with Interferon and Ribavirin include flu-like symptoms mostly due to interferon, cytopenias and haemolysis induced by Ribavirin. Psychiatric changes due to interferon, occur in up to 50% and thyroid abnormalities requiring therapy occur in about 1 to 5% treated with interferon. Autoimmune disease and retinal haemorrhages have also been reported. In addition, combination therapy is associated with significant risks in patients with renal dysfunction, cardiac disease and haemolytic anaemias as treatment may be associated with anaemia. Patients who are depressed or suicidal should also be excluded (2).

To this point little DNA microarray work done has been done with HCV. However, what work has been done is interesting and shows promise. In studies comparing Hepatitis B (HBV) with Hepatitis C, HBV infection was found to express genes predominantly involved in inflammation. In contrast, with HCV infection anti-inflammatory genes were found to be expressed (3). In another study HCV associated cirrhosis has been shown to be characterized by proinflammatory, pro-fibrotic and proapoptotic gene expression profiles (4).

The progression of HCV infection by gene expression analysis of liver biopsies in acutely infected chimpanzees that develop persistent infection, transient viral clearance, or sustained clearance has been examined. Transient and sustained viral clearance were uniquely associated with induction of IFN-gamma-induced genes and other genes involved in antigen processing and presentation and the adaptive immune response. The study revealed genome-wide transcriptional changes that reflect the establishment, spread, and control of infection, and they reveal potentially unique antiviral programs associated with clearance of HCV infection (5).

In-vitro studies in the human cell line Huh7 has shown that on exposure of the cells to Interferon 50 genes were up-regulated by at least twofold in control clones, whereas induction of 9 of the 50 genes was significantly reduced in those Huh7 clones expressing NS5A. Interferon-alpha activity has been found to be inhibited by the HCV protein NS5A. The strongest effect of NS5A on Interferon response was observed on the OAS-p69 gene with reduced expression. In addition, Huh7 cells expressing NS5A showed an up-regulation of interleukin-8 a proinflammatory cytokine. As a result this study postulated a mechanism for NS5A mediated interferon resistance (6).

In a recent study microarray gene profiling of peripheral blood mononuclear cells from hepatitis C patients treated with Interferon-alpha was performed. 88 genes directly relating to functions of immune cells were up-regulated, including genes involved in antigen processing and presentation, T-cell activation, lymphocyte trafficking, and effector functions, suggesting that Interferon-alpha up-regulates multiple genes involving different aspects of immune responses to enhance immunity against hepatitis C virus (7).

Currently, treatment for HCV still has a significant non-responder rate and is associated with side effects which limits many individuals from receiving treatment. Already molecular profiling by DNA microarrays has identified potential genetic targets which may have a role in the pathogenesis of HCV-associated hepatitis and more importantly possible targets which have a role in response to Interferon treatment. The work proposed here hopes to build on this body of knowledge and may lead to improved treatment modalities for HCV.

Methods/Experimental Design:

Approval from the Alfred Hospital Ethics Committee will be obtained and subjects will be recruited via the Alfred Hospital's Hepatitis Clinics. Informed consent for the study will be obtained after its purpose is explained verbally and via a plain English statement. Informed consent will also include consent for liver biopsies. Initially, a pilot study will be undertaken in which only one subject will be recruited to both the experimental and control arm of the study. Once the results from this pilot study have been analysed the study will be expanded to encompass a greater number of individuals.

Liver biopsies will be performed on the following groups.

1. HCV positive patients prior to commencement and at the end of treatment with either standard or pegylated Interferon plus Ribavirin. This group will be subdivided into responders and non-responders to treatment. Core liver biopsies under ultra-sound guidance are already routinely performed on this group prior to the commencement of treatment. For the purpose of this study non-responders to combination therapy are those individuals who remain HCV-RNA positive at the end of treatment.
2. Control population consisting of patients undergoing laparotomy for diseases not involving the liver. These biopsies would be obtained at the time of surgery.

Enough liver tissue (approximately 1-2 mg) will be obtained to isolate messenger RNA (mRNA) by oligo dT chromatography. Once isolated the mRNA will be reverse transcribed to complementary DNA (cDNA). This cDNA will then be labeled with a fluorescent reporter molecule. Hybridization of the labeled liver cDNA will then occur with the DNA microarray. It is envisaged that the microarray will be commercially obtained and consist of human cDNA. There is enough DNA on the microarray that two lots of labeled liver cDNA with different fluorescent markers (i.e. red and green) can be hybridized to the array at the same time without any interference. The following hybridizations would then be set up.

Reporter molecule 1: HCV +ve group. cDNA Reporter molecule 2: HCV -ve group. cDNA

Hybridization 1 Responder to Rx. Before Rx Control cDNA

Hybridization 2 Responder to Rx. After Rx Control cDNA

Hybridization 3 Non responder to Rx. Before Rx Control cDNA

Hybridization 4 Non responder to Rx. After Rx Control cDNA

Rx = treatment.

The hybridized array will then be scanned and commercially available software packages will be used to help in the interpretation of the results (8). Genes or groups of genes of particular interest include:

1. Pro-inflammatory response genes

   * Th-1 cytokines such as Gamma Interferon (IFN), Interleukin-2 (IL-2) and Tumour Necrosis Factor-beta (TNF-ß). Th1 cytokines promote production of opsonizing antibodies (e.g., IgG1) and induction of cellular cytotoxicity and macrophage activation. Th1 responses are prominent in the defence against pathogens which replicate intracellularly.
   * Tumour Necrosis Factor (TNF) and TNF receptor family of molecules which are strongly pro-inflammatory and involved in immune regulation.
   * Interleukin-12 (IL-12) which is a key cytokine that protects the host from viral and microbial infection. It links the innate and acquired arms of the immune system.
   * Interleukin-18 (IL-18) which has been shown to act as a chemoattractant.
2. Genes involved in a pro-fibrotic response.

   * Transforming growth factor beta (TGFbeta) which causes fibroblast proliferation.
   * Procollagen I and II.
   * Platelet-derived growth factor (PDGF) and PDGF beta receptor over-expression have been linked to development of fibrotic disease as well as cancer and atherosclerosis.
   * Matrix metalloproteinases play a pivotal role in angiogenesis and have a role in tumorigenesis.
   * Fibroblast Growth Factor.
   * Vascular Endothelial Growth Factor (VEGF) which is known for its angiogenic properties.
   * Connective tissue growth factor which stimulates collagen production.

In addition, novel genes previously unidentified, with differential expression will be looked for and will be characterized.

References relevant to this project (from literature search)

1. Chopra, S. Treatment of chronic hepatitis C infection: Recommendations. In: Up To Date, Rose, BR(Ed), Up To Date, Wellesley. MA, 2002.
2. Bonis, PLA, Chopra, S. Administration of combined interferon alfa-2b and ribavirin in the treatment of hepatitis C infection. In: Up To Date, Rose, BR(Ed), Up To Date, Wellesley. MA, 2002.
3. Honda, M, Kaneko, S, Kawai, H, et al. Differential gene expression between chronic hepatitis B and C hepatic lesions. Gastroenterology 2001; 120: 955-66.
4. Shackel, NA, McGuinness, PH, Abbott, CA, et al. Insights into the pathobiology of hepatitis C virus-associated cirrhosis: analysis of intrahepatic differential gene expression. Am J Pathol 2002; 160: 641-54.
5. Su, AI, Pezacki, JP, Wodicka L, et al. Genomic analysis of the host response to hepatitis C virus infection. Proc Natl Acad Sci 2002;99:15669-74.
6. Girard, S, Shalhoub, P, Lescure, P, et al. An altered cellular response to interferon and up-regulation of interleukin-8 induced by the hepatitis C viral protein NS5A uncovered by microarray analysis. Virology 2002; 295: 272-83.
7. Ji, X, Cheung, R, Cooper, S, et al.Interferon alfa regulated gene expression in patients initiating interferon treatment for chronic hepatitis C. Hepatology 2003;37:610-21.
8. Jenkins, RE, Pennington, SR. arrays for protein expression profiling: towards a viable alternative to two-dimensional gel electrophoresis. Proteomics 2001; 1: 12-29.

ELIGIBILITY:
Inclusion Criteria:

* HCV mono-infection, no coagulopathy and having a liver biopsy for consideration of treatment

Exclusion Criteria:

* Infection with HIV or HBV, excess ethanol (EtOH) consumption and other diseases of the liver

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-02; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Berzsenyi, MBBS, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia